CLINICAL TRIAL: NCT01224184
Title: Adapting the Women's CoOp for At-Risk Teens
Brief Title: Young Women's CoOp Study
Acronym: YWC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5UR6PS000665-04 (NIH)
Record Dates: First submitted 2010-10-13; First posted 2010-10-19 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: HIV; Sexual Risk; Sexually Transmitted Diseases; Substance Abuse; Violence; Victimization
Keywords: HIV; Sexually Transmitted Diseases; Substance Abuse Detection; Randomized Controlled Trial
MeSH Terms: conditions — Sexually Transmitted Diseases; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition (Active Comparator): Participants in this group will participate in three individual sessions and one group session of the nutrition intervention about healthy eating, physical activity and general wellness.
  Interventions: Behavioral: Staying Healthy and Eating Well
- Young Women's (Experimental): Participants in this group will participate in three individual sessions and one group session of the young woman-focused intervention about HIV/STIs, pregnancy, alcohol and other drug use, violence, gangs and other issues. This intervention is an adaptation of the evidence-based Women's CoOp (Principal Investigator (PI): Dr. Wendee M. Wechsberg).
  Interventions: Behavioral: Young Women's CoOp

INTERVENTIONS:
Behavioral: Young Women's CoOp — Participants in this group will participate in three individual sessions and one group session of the young woman-focused intervention about HIV/STIs, pregnancy, alcohol and other drug use, violence, gangs and other issues. This intervention is an adaptation of the evidence-based Women's CoOp (PI: Dr. Wendee M. Wechsberg).
  Arms: Young Women's
Behavioral: Staying Healthy and Eating Well — Participants in this group will participate in three individual sessions and one group session of the nutrition intervention about healthy eating, physical activity and general wellness.
  Arms: Nutrition

SUMMARY:
The purpose of this study is to test the efficacy of a cultural-, age- and gender-focused Human Immunodeficiency Virus (HIV) prevention intervention in reducing risk behaviors among African-American young women relative to general health intervention.

DETAILED DESCRIPTION:
This study completed an extensive formative phase to adapt the Women's CoOp intervention to specifically address the needs of young out-of-school adolescent African-American females with regard to knowledge about sexually transmitted infections (STIs), HIV and sexuality, health consequences of substance abuse, relationships with males, condom communication and social support, and HIV risk-reduction and violence prevention methods. During this phase, in-depth interviews, focus groups, pretesting and pilot testing were conducted to adapt and refine the intervention for the clinical trial.

The aim of this trial is to:

• Evaluate the efficacy of the cultural-, age-, and gender-focused intervention (Young Women's CoOp) relative to an equal attention control nutrition intervention in terms of changes in behaviors (e.g., condom use, substance use, violence prevention).

At study enrollment/baseline, participants completed a questionnaire and baseline drug and pregnancy testing, and were randomized into one of two programs: Young Women's CoOp or Staying Healthy and Eating Well (Nutrition)-both which included 3 individual intervention sessions and 1 group activity. Follow-ups were conducted 3-months post-intervention and 6-months post-intervention and included a questionnaire and drug testing.

The study has since been completed and analysis and manuscript preparation is underway. Two abstracts have been accepted to American Public Health Association conferences in 2012 and 2013. The five papers in progress or published include:

1. Efficacy of the Young Women's Coop - analysis complete, manuscript being drafted
2. Summary of qualitative findings from interviews and focus groups - published September 2013
3. Homelessness and abuse- in final preparation
4. Correlates of gang affiliation - manuscript complete, CDC clearance obtained, under review.
5. Post intervention social determinants - re-analyses and re-write

ELIGIBILITY:
Inclusion Criteria:

* Female
* Black/African-American
* 16-19 years of age
* Have dropped out of school at least once or are having problems that they have considered dropping out of school, and have not yet completed high school or GED program
* Have not graduated from a high school or alternative school, or completed a General Education Development (GED) program
* Have had vaginal sex at least once in the past 90 days with a male partner
* Have used one of the following at least once in the past 90 days--alcohol, marijuana, cocaine/crack, heroin, ecstasy, methamphetamine, any prescription drugs not prescribed to them, or any other illicit substance.
* Will be in the area for the next 8 months
* Has not participated in previous formative activities of the study (e.g., interviews, focus groups, pretesting and pilot testing),

Exclusion Criteria:

* Not interested in coming to a health behavior study
* Not able to attend 4 sessions and 2 follow ups

Ages: 16 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 237 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes in behaviors, including condom use, substance use and violence prevention | 3, and 6- months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (2):
- United States (2):
  - RTI International; Substance Abuse Treatment Evaluations and Interventions (SATEI) Community-Based Field Site - Durham, Durham, North Carolina
  - RTI International - Headquarters, Research Triangle Park, North Carolina

REFERENCES:
- [Background] Wechsberg WM, Browne FA, Ellerson RM, Zule WA. Adapting the evidence-based Women's CoOp intervention to prevent human immunodeficiency virus infection in North Carolina and international settings. N C Med J. 2010 Sep-Oct;71(5):477-81. No abstract available. PMID 21473554
- [Background] Browne, F. A., Wechsberg, W. M., White, V. L., Middlesteadt Ellerson, R., Raiford, R. L., Carry, M. G., Herbst, J.H. (in press).